CLINICAL TRIAL: NCT04677595
Title: A Phase II, Multicenter, Two-cohort Study of Oral MET Inhibitor Capmatinib in Chinese Adult Patients With EGFR Wild-type (wt), ALK Rearrangement Negative, MET Exon 14 Skipping Mutations, Advanced Non-small Cell Lung Cancer (NSCLC) Who Are Treatment Naive or Failed One or Two Prior Lines of Systemic Therapy
Brief Title: Study of Capmatinib in Chinese Adult Patients With Advanced Non-small Cell Lung Cancer Harboring MET Exon 14 Skipping Mutation
Acronym: GeoMETry-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2204
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non small cell lung cancer; Non small cell carcinoma; INC280; capmatinib; NSCLC; MET mutation; MET exon14; EGFTwt; ALK negative; Epidermal growth factor receptor wild type
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Treatment Naive participants
  Interventions: Drug: Capmatinib
- Cohort 2 (Experimental): Participants received one or two prior lines of treatment
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — 400 mg of capmatinib tablets, administered orally twice daily
  Other Names: INC280

SUMMARY:
The purpose of the study is to learn whether the study treatment (capmatinib), which already shows efficacy and safety in non-Chinese patients, could help Chinese patients with controlling their lung cancer in a safe way. Participants will have a type of lung cancer called non-small cell lung lancer (NSCLC), with a specific alteration in a part of their DNA (called mutation) of the MET gene, within a specific part of this gene called exon 14.

Participants who have advanced (or metastatic) non-small cell lung cancer with specific mutations in the MET gene but without mutations in the EGFR or ALK genes, who are aged 18 years or older will be enrolled in this study.

The study drug, capmatinib (also known as INC280), is an oral drug that is called a 'targeted' medicine, which means it targets particular processes that may not be working properly in cancer cells (called dysregulation). The dysregulation of the MET signaling in cancer cells of patients with NSCLC is believed to make the cancer worse. Capmatinib has been shown to selectively block the effects of the MET gene and therefore may help in keeping the disease under control, stopping cancer cells from growing.

DETAILED DESCRIPTION:
This is an open-label, multicenter two-cohort phase II study. Chinese adult participants with EGFR wild-type (wt) (EGFR mutations that predict sensitivity to EGFR therapy, including, but not limited to exon 19 deletions and exon 21 L858R substitution mutations), anaplastic lymphoma kinase (ALK) rearrangement negative, advanced (stage IIIB, IIIC or IV) NSCLC disease harboring MET exon 14-skipping (METΔex14) mutations as determined by a Novartis central molecular laboratory will be treated in this study. Cohort 1 will include treatment naive participants and Cohort 2 participants who failed one or two prior lines of therapy in the advanced stage (stage IIIB, IIIC or IV). Each participant will receive 400 mg capmatinib tablet twice daily (BID).

The primary endpoint is the overall response rate (ORR) by cohort as per the blinded independent review committee (BIRC) review. ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR) according to RECIST 1.1.

The primary analysis will be performed using full analysis set (FAS). The primary efficacy endpoint ORR will be estimated and the exact 95% confidence interval (CI) will be provided by cohort.

ELIGIBILITY:
Key Inclusion Criteria:

* Chinese adult ≥ 18 years old at the time of informed consent
* Histologically confirmed stage IIIB, IIIC or IV NSCLC at the time of study entry, not amenable to curative surgery or radiation or multi-modality therapy (according to staging definition in CSCO guidelines for primary lung cancer, 2019).
* Histologically or cytologically confirmed diagnosis of NSCLC that is:

  1. EGFR wt: The EGFR wt status assessed as part of standard of care (EGFR mutations that predict sensitivity to EGFR therapy, including, but not limited to exon 19 deletions and exon 21 L858R substitution mutations)
  2. AND ALK rearrangement negative: assessed as part of standard of care by validated test
  3. AND either:

Cohort 1: Treatment naive participants with MET mutations, or Cohort 2: Pre-treated participants with MET mutations

* Cohort 1: participants must not have received any systemic therapy for advanced/metastatic disease (stage IIIB, IIIC or IV NSCLC). Neo-adjuvant and adjuvant systemic therapies will not count as one prior line of treatment if relapse occurred > 12 months from the end of the neo-adjuvant or adjuvant systemic therapy.
* Cohort 2: participants must have failed one or two prior lines of systemic therapy for advanced/metastatic disease (stage IIIB, IIIC or IV NSCLC).
* At least one measurable lesion according to RECIST v1.1.
* Adequate organ function
* ECOG performance status (PS) ≤1

Key Exclusion Criteria:

* Prior treatment with any MET inhibitor or HGF-targeting therapy.
* Known druggable molecular alterations (such as ROS1 translocation or BRAF mutation, etc.) which might be a candidate for alternative targeted therapies as applicable per local regulations and treatment guidelines.
* Participants with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Presence or history of interstitial lung disease or interstitial pneumonitis, including, clinically significant radiation pneumonitis affecting activities of daily living or requiring therapeutic intervention.
* Substance abuse, active infection (including active hepatitis B and C, participants whose disease is controlled under antiviral therapy are eligible, and human immunodeficiency virus (HIV) history positive) or other severe, acute, or chronic medical or psychotic conditions or laboratory abnormalities that in the opinion of the investigator may increase the risk associated with study participation, or that may interfere with the interpretation of study results.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) by blinded independent review committee (BIRC) assessment, by cohort | Up to approximately 23 months
  ORR is defined as the proportion of participants with a best overall response (BOR) defined as complete response or partial response (CR+PR) by BIRC assessment per RECIST 1.1

SECONDARY OUTCOMES:
Duration of response (DOR) as assessed by BIRC, by cohort | From first documented response to first documented progression or death due to any cause, whichever comes first, assessed up to approximately 23 months
  DOR, calculated as the time from the date of the first documented CR or PR by BIRC per RECIST 1.1 to the first documented progression or death due to any cause for participants with PR or CR
Overall response rate (ORR) and duration of response (DOR) by investigator assessment, by cohort | Up to approximately 23 months
  ORR (CR+PR) and DOR per RECIST 1.1 by investigator assessment
Time to response (TTR) by investigator and by BIRC assessment, by cohort | From first dose to first documented response of either CR or PR, assessed up to approximately 23 months
  TTR, calculated as the time from first dose of capmatinib to first documented response (CR+PR) for participants with PR or CR per RECIST 1.1 by BIRC and investigator
Disease Control Rate (DCR) by investigator and by BIRC assessment, by cohort | Up to approximately 23 months
  DCR, calculated as the proportion of participants with BOR of CR, PR, or SD (stable disease) per RECIST 1.1 by BIRC and investigator
Progression Free Survival (PFS) by investigator and by BIRC assessment, by cohort | From first dose to the date of first documented progression or death from any cause, whichever comes first, assessed up to approximately 23 months
  PFS, defined as time from first dose of capmatinib to progression or death due to any cause per RECIST 1.1 by BIRC and investigator
Overall survival (OS) | From first dose to death due to any cause, assessed up to approximately 42 months
  OS is defined as the time from first dose to the date of death due to any cause.
Overall intracranial response rate (OIRR) | Up to approximately 23 months
  Overall intracranial response rate (OIRR) calculated as the proportion of participants with a confirmed best overall intracranial response (BOIR) of CR or PR per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria as assessed by BIRC
Intracranial disease control rate (IDCR) | Up to approximately 23 months
  Intracranial disease control rate (IDCR), defined as the proportion of participants with a confirmed BOIR of CR or PR or SD (or non-CR/non-Progressive Disease) per RANO-BM criteria as assessed by BIRC review.
Time to intracranial response (TTIR) | Up to approximately 23 months
  Time to intracranial response (TTIR) defined as the time from the date of the start of study treatment to the date of the first documented intracranial response of either CR or PR per RANO-BM criteria as assessed by BIRC
Duration of intracranial response (DOIR) | Up to approximately 23 months
  Duration of intracranial response (DOIR) defined as the time from the date of first documented intracranial response of either CR or PR to the date of the first documented intracranial progression per RANO-BM criteria as assessed by BIRC review or date of death due to any cause.
Association between MET mutation status as measured in ctDNA at baseline with capmatinib efficacy | Up to approximately 23 months
  ORR, DOR and PFS per RECIST 1.1 for participants by MET mutation status assessed in circulating tumor DNA (ctDNA) at baseline, both by BIRC and investigator. The association between MET mutation status as measured in ctDNA at baseline with ORR, DOR and PFS will be established using Kaplan-Meier curve by cohort separately. Median survival together with their 95% confidence intervals will be reported.
Plasma capmatinib concentration | Cycle 2 Day 1 pre-dose, 0.5-1.5 hours post-dose and 3-5 hours post dose and Cycle 3 Day 1 pre-dose. Each cycle duration is 21 days
  Steady state Ctrough and steady state 0.5- 1.5 hour and 3-5 hours post-dose concentrations
Change from baseline in score as per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Cycle 1 Day 1, Cycle 3 Day 1 and then every 6 weeks up to approximately 23 months. Each cycle duration is 21 days.
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients.
Change from baseline in score as per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Lung Cancer Module (QLQ-LC13) | Cycle 1 Day 1, Cycle 3 Day 1 and then every 6 weeks up to approximately 23 months. Each cycle duration is 21 days.
  EORTC QLQ-LC13 is a 13-item lung cancer specific questionnaire.
Change from baseline in score as per European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) questionnaire | Cycle 1 Day 1, Cycle 3 Day 1 and then every 6 weeks up to approximately 23 months. Each cycle duration is 21 days.
  EQ-5D-5L is a standardized measure to assess the overall health-related quality of life in patients.
Time to deterioration in symptoms of brain metastases, with the NCCN FACT-Brain Symptom Index symptom module (FBrSI) | Cycle 1 Day 1, Cycle 3 Day 1 and then every 6 weeks up to approximately 23 months. Each cycle duration is 21 days.
  National Comprehensive Cancer Network Functional Assessment of Cancer Therapy (NCCN FACT) - Brain Symptom Index version 2.0 (FBrSI) symptom module, consisting of 24 items with a recall period of the past 7 days, will explore changes in symptoms associated with potential brain metastases.

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Novartis Investigative Site, Xiamen, Fujian
  - Novartis Investigative Site, Foshan, Guangdong
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.